CLINICAL TRIAL: NCT05219734
Title: MRD Assay Evaluates Recurrence and Response Via a Tumor Informed Assessment
Acronym: MARIA
Status: Active, not recruiting | Type: Observational
Sponsor: Invitae Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: CR-001-016
Record Dates: First submitted 2021-12-20; First posted 2022-02-02 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Cancer; Solid Tumor; Non Small Cell Lung Cancer; Colorectal Cancer; Bladder Cancer
Keywords: minimal residual disease; MRD; ctDNA; circulating tumor DNA
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Urinary Bladder Neoplasms; Neoplasm, Residual

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples type to be collected is blood.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Personalized Cancer Monitoring (PCM) — personalized molecular test for solid tumor cancer patients that may detect the presence of circulating tumor DNA (ctDNA) and molecular residual disease (MRD), also known as minimal residual disease

SUMMARY:
This study recruits patient with solid tumor types for sample collection and monitoring. Participants will provide blood and archival tissue samples in order to create a Personalized Cancer Monitoring (PCM) assay. This assay will be used to detect circulating tumor DNA (ctDNA) levels in the blood over time and hopefully contribute to improvements in residual disease detection methods for future patients.

Results from this assay will be provided to participants and providers but providers are not asked to change patient care based on this information.

DETAILED DESCRIPTION:
This study involves collection of tumor tissue (from a standard biopsy and/or surgery) as well as blood samples over time in order to allow the creation of a Personalized Cancer Monitoring (PCM) assay. Additional blood samples are taken throughout the patient's treatment and follow-up period.

Each participant will submit one blood sample when they begin participation in the research study. Participants will be asked to submit follow up samples several times per year (annually, at minimum), with the exact frequency varying by stage and type of cancer. In general, participants will not be asked to come into the clinic more frequently than their already needed clinic visits.

If the cancer-specific mutations identified by the PCM are detected in the blood samples provided as part of the study, this may would suggests that residual cancer may be present. This is an observational study comparing MRD results to standard of care methods and collecting provider and patient perspectives, using surveys. Physicians will be informed of all PCM results in the form of a clinical report. Physicians are not asked to base treatment decisions on these results.

ELIGIBILITY:
Inclusion Criteria

1. Stated ability to give informed consent by participant.
2. Stated health status of participant as healthy enough to provide Biological Material.
3. Individuals diagnosed with solid cancer of any type, including but not limited to colorectal, non-small cell lung, breast, ovarian and bladder cancers, regardless of the length of time since diagnosis and regardless of previous therapies.
4. Participant is of any biological sex and >18 years of age
5. Participant has not undergone a blood transfusion within the previous three weeks

Exclusion Criteria

1. Participants who are deemed medically unstable
2. Participants who are deemed to be "difficult to draw" blood from.
3. Participants who are <18 years of age
4. Participants diagnosed with CNS cancers, sarcomas or hematologic malignancies such as leukemia or lymphoma .
5. Participants with more than one primary cancer
6. Participants with FFPE slides older than 10 years
7. Participants who are pregnant
8. Any other reason that, in the Investigator's judgment, that would preclude the participant from being able to participate in the study
9. Participants for which a pathology report is not available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study seeks to enroll patients of all solid tumor types across many clinical sites with emphasis on early stage non-metastatic Colorectal, Non small cell lung cancer, breast, ovarian and bladder cancers.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-11-29 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Through study completion, up to 5 years
Relapse Free Survival | Measured through study completion, assessed yearly up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Ed Esplin, MD, PhD, Study Director — Invitae Corporation; Michael Korn, Study Director — Invitae Corporation
Locations (2):
- United States (2):
  - Columbus Regional Health, Columbus, Indiana
  - Onslow Radiation, Jacksonville, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
Invitae may share de-identified information and data generated through the study with third parties, including biopharmaceutical companies and biomedical researchers (e.g. academic), for clinical trials, drug development, and other disease-related research purposes.
  Only a subset of Invitae personnel will have access to PHI. The PHI will be stored in a secure location and will only be made available to Invitae personnel involved in the Study. Any academic publication of data analysis from this Study will use de-identified information only.